CLINICAL TRIAL: NCT03196544
Title: Novel Behavioral Intervention to Target Social Reward Sensitivity and Attachment
Brief Title: Novel Behavioral Intervention to Enhance Social Connections in Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Charles Taylor, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 140102
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Anxiety Disorders and Symptoms; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social Approach Training (5 sessions) (Experimental)
  Interventions: Behavioral: Social Approach Training (5 sessions)
- Social Approach Training (10 sessions) (Experimental)
  Interventions: Behavioral: Social Approach Training (10 sessions)
- Delayed Treatment (Waitlist) (No Intervention)

INTERVENTIONS:
Behavioral: Social Approach Training (5 sessions) — 5 one-hour, clinician-administered treatment sessions focused on presenting rationale and instructions for completing positive activity exercises (e.g., gratitude, acts of kindness) designed to increase positive emotions, cognitions, and behaviors.
  Arms: Social Approach Training (5 sessions)
Behavioral: Social Approach Training (10 sessions) — 10 one-hour, clinician-administered treatment sessions focused on presenting rationale and instructions for completing positive activity exercises (e.g., gratitude, acts of kindness) designed to increase positive emotions, cognitions, and behaviors.
  Arms: Social Approach Training (10 sessions)

SUMMARY:
The overall goal of this project is to develop a novel transdiagnostic behavioral treatment -- social approach training -- intended to enhance positive social connections in individuals with elevated anxiety and/or depression. Social relationship impairments are pervasive and debilitating consequences of anxiety and depression. Existing treatments have some beneficial impact on social functioning; however, many people continue to have few and/or poor quality relationships following treatment, even after experiencing symptom relief. This study will evaluate the effects of social approach training on the brain systems that have been shown to be important for establishing positive connections with others. Approximately 60 individuals (ages 18-55) seeking treatment for anxiety or depression will participate in this study. Participants will be randomly assigned with equal probability to one of two versions of social approach training (5 or 10 sessions) or a waitlist (assessment only) control group. Participants will be assessed at baseline and post-treatment and compared on measures assessing brain responses to social reward (primary outcome), as well as physiological, behavioral, and emotional responses to social reward (secondary outcomes). It is hypothesized that participants assigned to social approach training will display greater increases from pre- to post-treatment in activity in brain systems that regulate the processing of social reward (e.g., striatum) relative to participants in the control group. This study will also determine whether the 5- vs. 10-session versions of the treatment program result in meaningful differences, compared to each other, in how the brain responds to social reward.

ELIGIBILITY:
Inclusion Criteria:

1. Score on the PHQ-9 is 10 or higher and/or score on the OASIS is 8 or higher.
2. Social Connectedness Scale Revised (SCSR) < 90
3. Sheehan Disability Scale (SDS) - Social Domain ≥ 5
4. Between the ages of 18-55, inclusive.
5. Have sufficient proficiency in English language to understand and complete interviews, questionnaires, and all other study procedures.

Exclusion Criteria:

1. No telephone or easy access to telephone.
2. Any substance use disorder in the past year except subjects with mild alcohol, nicotine, caffeine, and marijuana use disorders will be permitted in the study.
3. Bipolar I or Psychotic disorders.
4. Moderate to severe traumatic brain injury with evidence of neurological deficits, neurological disorders, or severe or unstable medical conditions that might be compromised by participation in the study.
5. Current and regular use (more days than not during the past 30 days) of a medication that could affect brain functioning, such as anxiolytics, antipsychotics, antidepressants, mood stabilizers, beta-blockers, sleep medications, opioids/codeine, migraine medications.
6. MRI contraindications including: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60 minutes; prior neurosurgery; tattoos with metal dyes, unwillingness to remove body piercings, and pregnancy.
7. non-correctable vision or hearing problems, as some tests require intact sensory functioning.
8. Concurrent psychosocial treatment: Participants completing ongoing empirically supported psychosocial treatment for the presenting problem will be required to meet 12-week stability criteria so that symptom changes as a result of other psychosocial treatments are not confounded with changes due to the research.
9. Inability to complete the initial assessment battery or treatment sessions.
10. Clinical conditions assessed by the interviewer that necessitate more imminent clinical care (e.g., active suicidal ideation): These criteria are in place so participants with these other, more several symptoms can be referred for appropriate mental health services.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in neural activation during social reward processing | Baseline, 10 weeks
  Change from pre- to post-assessment in neural activation measured using functional magnetic resonance imaging (fMRI) during reward trials of the social incentive delay (SID) task

SECONDARY OUTCOMES:
Change from baseline in response to a social interaction task | Baseline, 10 weeks
  Change from pre- to post-assessment in physiology, behavior, motivation, and affect in response to a social interaction task

OTHER OUTCOMES:
Change from baseline in social functioning as measured by the NIH Toolbox Companionship Friendship survey | Baseline, 10 weeks
  NIH Toolbox Companionship Friendship survey measures social functioning. Items are answered on a 5 point scale, 1 (Never) to 5 (Always). The NIH Toolbox Companionship Friendship survey ranges from 8-40 and higher scores indicate greater perceived availability of friends or companions with whom to interact or affiliate.
Change from baseline in social functioning as measured by the NIH Toolbox Loneliness Surveys | Baseline, 10 weeks
  The NIH Toolbox Loneliness survey measures social functioning. Items are answered on a 5 point scale, 1 (Never) to 5 (Always). The NIH Toolbox Loneliness survey ranges from 5-25 and higher scores indicate greater social isolation and feelings of loneliness.
Change from baseline in social functioning as measured by the Social Network Survey | Baseline, 10 weeks
  The Social Network Survey measures social functioning by looking at the size and density of a participants social network. Higher scores indicate greater levels of social functioning.
Change from baseline in social connectedness as measured by the Social Connectedness Scale Revised (SCSR) | Baseline, 10 weeks
  The SCSR measures social connectedness. Items are answered on a 6 point scale, 1 (Strongly disagree) to 6 (Strongly agree). The SCSR ranges from 20-120 and higher scores indicate greater levels of social connectedness.
Change from baseline in positive affect as measured by PROMIS Positive Affect - Short Form 15a survey | Baseline, 10 weeks
  The PROMIS Positive Affect - Short Form 15a survey measures positive affect. Items are answered in a 5 point scale, 1 (Not at all) to 5 (Very much). The PROMIS Positive Affect - Short Form 15a survey ranges from 15-75 and higher scores indicate higher levels of positive affect.
Change from baseline in positive affect as measured by Positive and Negative Affect Schedule | Baseline, 10 weeks
  The Positive and Negative Affect Schedule (PANAS) measures positive affect. Items are answered on a 5 point scale, 1 (Very slightly or not at all) to 5 (Extremely). The positive affect scale ranges from 10-50 and higher scores indicate greater levels of positive affect.
Change from baseline in positive affect as measured by Modified Differential Emotions Scale | Baseline, 10 weeks
  The Modified Differential Emotions Scale (mDES) measures positive emotions. Items are answered on a 5 point scale, 0 (Never/Not at all) to 4 (Most of the time/Extremely). Higher scores on the positive emotions sub-scale indicate higher levels of positive emotion.
Change from baseline in psychological well-being as measured by PROMIS General Life Satisfaction - Short Form 5a survey | Baseline, 10 weeks
  The PROMIS General Life Satisfaction - Short Form 5a survey measures psychological well-being. The PROMIS General Life Satisfaction items are answered on a 7 point scale, 1 (Strongly disagree) to 7 (Strongly agree). The PROMIS General Life Satisfaction survey ranges from 5-25 and higher scores indicate higher levels of life satisfaction.
Change from baseline in psychological well-being as measured by PROMIS Meaning and Purpose - Short Form 6a survey | Baseline, 10 weeks
  The PROMIS Meaning and Purpose - Short Form 6a survey measure psychological well-being. The PROMIS Meaning and Purpose items are answered on a 5 point scale, 1 (Not at all) to 5 (Very much). The PROMIS Meaning and Purpose survey ranges from 6-30 and higher scores indicate higher levels of self reported meaning and purpose in ones life.
Change from baseline in negative affect as measured by the Positive and Negative Affect Schedule | Baseline, 10 weeks
  The Positive and Negative Affect Schedule (PANAS) measures negative affect. Items are answered on a 5 point scale, 1 (Very slightly or not at all) to 5 (Extremely). The negative affect scale ranges from 10-50 and lower scores indicate lower levels of negative affect.
Change from baseline in negative affect as measured by the Modified Differential Emotions Scale | Baseline, 10 weeks
  The Modified Differential Emotions Scale (mDES) measures negative emotions. Items are answered on a 5 point scale, 0 (Never/Not at all) to 4 (Most of the time/Extremely). Lower scores on the negative emotions sub-scale indicate lower levels of negative emotion.
Change from baseline in anxiety as measured by PROMIS Anxiety 7a survey | Baseline, 10 weeks
  The PROMIS Anxiety 7a survey measures symptoms of anxiety. Items are rated on a 5 point scale, 1 (Never) to 5 (Always). The scale ranges from 7-35 and higher scores indicate higher levels of anxiety.
Change from baseline in anxiety as measured by the Overall Anxiety Severity and Impairment Scale | Baseline, 10 weeks
  The Overall Anxiety Severity and Impairment Scale (OASIS) measures frequency, severity, and functional impairment of anxiety symptoms. Items are rated on a 4 point scale, 0 (None) to 4 (Extreme). The scale ranges from 0-20 and higher scores indicate higher levels of anxiety.
Change from baseline in depression as measured by PROMIS Depression 8b survey | Baseline, 10 weeks
  The PROMIS Depression 8b survey measures symptoms of depression. Items are rated on a 5 point scale, 1 (Never) to 5 (Always). The scale ranges from 8-45 and higher scores indicate higher levels of depression.
Change from baseline in depression as measured by the Patient Health Questionnaire-9 | Baseline, 10 weeks
  The Patient Health Questionnaire-9 (PHQ-9) measures depression symptoms. Items are rated on a 4 point scale, 0 (Not at all) to 3 (Nearly every day). The scale ranges from 0-27 and higher scores indicate higher levels of depression.
Change from baseline in functional impairment as measured by the Sheehan Disability Scale | Baseline, 10 weeks
  The Sheehan Disability Scale measures functional impairment. Items are rated on a 11 point scale, 0 (Not at all) to 10 (Extremely). The scale ranges from 0-30 and higher scores indicate higher levels of functional impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Altman Clinical and Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Taylor CT, Lyubomirsky S, Stein MB. Upregulating the positive affect system in anxiety and depression: Outcomes of a positive activity intervention. Depress Anxiety. 2017 Mar;34(3):267-280. doi: 10.1002/da.22593. Epub 2017 Jan 6. PMID 28060463
- [Derived] Kryza-Lacombe M, Spaulding I, Ku CK, Pearson N, Stein MB, Taylor CT. Amplification of positivity for depression and anxiety: Neural prediction of treatment response. Behav Res Ther. 2024 Jul;178:104545. doi: 10.1016/j.brat.2024.104545. Epub 2024 Apr 23. PMID 38714105

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT03196544/Prot_ICF_000.pdf